CLINICAL TRIAL: NCT02615041
Title: The Pharmacodynamics of Meropenem in Patient With Ventilator-associated Pneumonia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sutep Jaruratanasirikul (Other)
Collaborators: Prince of Songkla University (Other)
Responsible Party: Sponsor-Investigator, Sutep Jaruratanasirikul, Principal Investigator, Prince of Songkla University
Organization: Prince of Songkla University (Other)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: MR-13/2545
Record Dates: First submitted 2015-11-24; First posted 2015-11-25 (Estimated); Last update posted 2015-11-25 (Estimated); Status verified 2015-11

CONDITIONS: Ventilator-Associated Pneumonia
Keywords: Meropenem; Ventilator-Associated Pneumonia; population pharmacokinetics; pharmacokinetics; pharmacodynamics
MeSH Terms: conditions — Pneumonia, Ventilator-Associated | interventions — Meropenem

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 g by bolus injection (Experimental): 1 g of meropenem with bolus injection every 8 h regimen
  Interventions: Drug: Meropenem
- 1 g by 3 h infusion (Experimental): 1 g of meropenem with 3 h infusion every 8 h regimen
  Interventions: Drug: Meropenem
- 2 g by 3 hinfusion (Experimental): 2 g of meropenem with 3 h infusion every 8 h regimen
  Interventions: Drug: Meropenem

INTERVENTIONS:
Drug: Meropenem — 1 g in 100 ml of normal saline solution and administered via bolus injection Blood samples (approximately 5 ml)will be obtained by direct venepuncture at the following time: before (time zero) and 10 and 30 min and 1, 1.5, 2, 2.5, 3.5, 4, 4.5, 5, 6, and 8 hh after 3rd dose of meropenem
  Other Names: Meronem
  Arms: 1 g by bolus injection
Drug: Meropenem — 1 g in 100 ml of normal saline solution and administered via an infusion pump at a constant flow rate over 3 h every 8 h.
  Blood samples (approximately 5 ml)will be obtained by direct venepuncture at the following time: before (time zero) and 10 and 30 min and
  1, 1.5, 2, 2.5, 3.5, 4, 4.5, 5, 6, and 8 h after the 3rd dose of meropenem.
  Other Names: Meronem
  Arms: 1 g by 3 h infusion
Drug: Meropenem — 2 g in 100 ml of normal saline solution and administered via an infusion pump at a constant flow rate over 3 h every 8 h.
  Blood samples (approximately 5 ml)will be obtained by direct venepuncture at the following time: before (time zero) and 10 and 30 min and 1, 1.5, 2, 2.5, 3.5, 4, 4.5, 5, 6, and 8 h after the 3rd dose of meropenem.
  Other Names: Meronem
  Arms: 2 g by 3 hinfusion

SUMMARY:
The study was a randomized three-way crossover study. Each subject received meropenem in three regimens at room temperature consecutively: (i) bolus injection of 1 g of meropenem over 10 min every 8 h for 24 h, (ii) 3-h infusion of 1 g of meropenem via an infusion pump at a constant flow rate every 8 h for 24 h, and(iii) 3-h infusion of 2 g of meropenem via an infusion pump at a constant flow rate every 8 h for 24 h.

Clinical and laboratory data such as Age,Sex, Body weight, Electrolyte, Vital signs, APACHE II score, BUN, Cr, Blood culture will be collected.

Nine patients will be enrolled in this study. After completion of the meropenem therapy for 3 days in this study, all patients will receive other sensitive antibiotics to eradicate their bacterial infections.

Meropenem pharmacokinetic studies were carried out during administration of the third dose of each regimen (16 to 24 h after the start of each regimen). Blood samples (approximately 5 ml) were obtained by direct venipuncture at the following times: before (time zero) and 10 and 30 min and

1, 1.5, 2, 2.5, 3.5, 4, 4.5, 5, 6, and 8 h after the third dose of each regimen.

The concentrations of meropenem were determined by reverse-phase high-performance liquid chromatography.

Concentration of meropenem in plasma will be simulated in Monte Carlo technique (Computer model) to get PK/PD index (40%T>MIC) and reported to % PTA(Probability Target Attainment) and %CFR (Cumulative Faction Response)

DETAILED DESCRIPTION:
Introduction:

Meropenem is a carbapenem antibacterial agent with a broad spectrum of activity against several pathogens. In common with other -lactams, the main pharmacokinetic/pharmacodynamic parameter that correlates with the therapeutic efficacy is the T>MIC, and administration by continuous infusion is the preferred route to maximize this parameter. However, in tropical countries the stability of meropenem is an important consideration when continuous infusion is to be used.

Objective:

The aim of this study was to demonstrate the T>MIC of meropenem when administered by a 3-h infusion compared with that when administered by bolus injection.

Study design:

The study was conducted with nine patients with ventilator-associated pneumonia. Each subject received meropenem in three regimens consecutively: (i) bolus injection of 1 g every 8 h for 24 h; (ii) 3-h infusion of 1 g every 8 h for 24 h; and (iii) 3-h infusion of 2 g every 8 h for 24 h.

Sample collections:

Meropenem pharmacokinetic studies were carried out during administration of the third dose of each regimen (16 to 24 h after the start of each regimen). Blood samples (approximately 5 ml) were obtained by direct venipuncture at the following times: before (time zero) and 10 and 30 min and 1, 1.5, 2, 2.5, 3.5, 4, 4.5, 5, 6, and 8 h after the third dose of each regimen.

Meropenem assay:

The concentrations of meropenem were determined by reverse-phase high-performance liquid chromatography. Cefepime (100 mcg/ml) was used as the internal standard, and the samples were extracted by the method of Ozkan et al.

Clinical data and pathogens collection:

1. Initial patient demographic data (age, sex, weight, diagnosis, APACHE II scores) will be collected upon enrollment in the study.
2. The Gram negative bacilli isolated from sputum in 9 patients will be collected and the MIC of the meropenem for pathogens will be determined by E tests upon enrollment in the study.

Duration of study:

Patients will receive meropenem for 3 days

Pharmacokinetic and pharmacodynamic analysis:

Concentration of meropenem in plasma will be simulated in Monte Carlo technique (Computer model) to get PK/PD index (40%T>MIC) and reported to % PTA (Probability Target Attainment) and %CFR (Cumulative Faction Response) Sample Size: Nine patients with VAP will be enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

* The patients were eligible for the study if they met the following criteria:

  1. older than 18 years
  2. clinical suspicion of VAP, defined by a new and persistent infiltrate on chest radiography associated with at least one of the following-purulent tracheal secretions, temperature of 38.3 celsius or higher, or a leukocyte count higher than 10000.

Exclusion Criteria:

* Patients were excluded from the study if they were pregnant or in circulatory shock (which was defined as a systolic blood pressure of 90 mmHg and poor tissue perfusion) or had documented hypersensitivity to meropenem or an estimated creatinine clearance(determined by the Cockcroft-Gault method) of 60 ml/min.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2004-01; Primary Completion 2005-01 (Actual); Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Concentration of meropenem in plasma | 8 hours profile after 3rd dose of meropenem
  Concentration of doripenem in plasma will be simulated in Monte Carlo technique (Computer model) to get PK/PD index (40%T>MIC) and reported to % PTA (Probability Target Attainment) and %CFR (Cumulative Faction Response).

CONTACTS AND LOCATIONS:
Overall Officials: Sutep Jaruratanasirikul, MD, Principal Investigator — Prince of Songkla University
Locations (1):
- Prince of Songkla University, Hat Yai, Changwat Songkhla, Thailand